CLINICAL TRIAL: NCT06590831
Title: Lactoferrin Alone ,Iron Alone Vs Lactoferrin Plus Iron for Treatment of Iron Deficiency Anemia During the 3rd Trimester of Pregnancy (Randomized Controlled Trial)
Brief Title: Lactoferrin Alone ,Iron Alone Vs Lactoferrin Plus Iron for Treatment of Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rehab Ahmed Amine
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-06

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: (lactoferrin Group) (Active Comparator): About 133 anemic pregnant women will be treated with lactoferrin only (pravotin 100mg ) twice daily for 4 weeks.
  Interventions: Drug: Lactoferrin
- Group B: (Amino acid chelated iron Group) (Active Comparator): About 133 anemic pregnant women will be treated with amino acid chelated iron only (phara fero 27) once daily for 4 weeks.
  Interventions: Drug: Lactoferrin
- Group C: (lactoferrin with amino acid chelated iron Group) (Active Comparator): About 133 anemic pregnant women will be treated with lactoferrin with amino acid chelated iron (phara fero 27 plus ) once daily for 4 weeks
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin — to compare between efficacy of lactoferrin alone and lactoferrin with iron for treatment of iron deficiency anemia during 3rd trimester of pregnancy
  Other Names: Iron

SUMMARY:
Iron deficiency (ID) and iron deficiency anemia (IDA) are the most common iron disorders throughout the world.

ID and IDA, particularly caused by increased iron requirements during pregnancy; represent a high risk for preterm delivery, fetal growth retardation, low birth weight, and inferior neonatal health. These pregnancy complications are thought to occur because of an increased iron requirement, related to enhanced blood volume and development of the fetoplacental unit.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines anemia in pregnancy as a hemoglobin (Hb) concentration of < 11 g/dl. Centers for disease control &prevention determine a cut of -off point 10.5 g/dl during 2nd trimester for diagnosis of IDA.

Iron deficiency anemia (IDA) is the most common type of anemia in pregnancy. The iron content of the body is normally kept constant by regulating the amount absorbed to balance the amount lost.

The WHO estimates that 46% of pregnant women in African region, 38% in Eastern Mediterranean region, 25% in European region and 24% in the region of the Americas are anemic mainly because of iron deficiency. Anemia is a common medical disorder affecting a lot of women in pregnancy in the developing countries.

Management of anemia remain an important issue in prenatal medicine. Correct diagnosis and treatment lead to effective management of fetal and maternal risk and improved prenatal outcome. Diet alone can't supply the 30-40 mg iron that is required for absorption of 4-6mg iron per day needed during the later stage of pregnancy so iron supplementation is strongly recommended for all females in developing countries.

Traditional therapeutic options of iron deficiency anemia during pregnancy were administration of oral iron shows lack of compliance and side effects and often limited intestinal absorption and bioavailability. The most used treatment for ID and IDA currently consists of oral administration of iron as ferrous sulphate. However, ferrous sulphate administration often fails to exert any significant effects on these pregnancy-associated pathologies, and frequently causes several adverse effects.

This is likely due to the poor bioavailability of inorganic iron requiring the administration of large quantity of ferrous sulphate. Lactoferrin is a multifunctional protein of the transferrin family. Lactoferrin is a globular glycoprotein with a molecular mass of about 80 kDa that is widely represented in various secretory fluids, such as milk, saliva, tears, and nasal secretions. Lactoferrin is also present in secondary granules of Polymorpho nuclear leucocyte and is secreted by some acinar cells. Lactoferrin can be purified from milk or produced recombinantly .

Lactoferrin (previously lactotransferrin)is a glycoprotein that belongs to transferrin family ,which includes protiens that may bind &transferrin.Lactoferrin levels in cow milk &human milk colostrum are roughly seven times higher than lactoferrin levels in milk prouduced later

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with single fetus
* All pregnant women in 3rd trimester (28w_36w) complaining of mild IDA
* Iron Deficiency Anemia mild anemia (hemoglobin level < 11 mg/dl , and serum ferritin level < 12 mg/dl).

Exclusion Criteria:

* Patients with a history of anemia due to any other causes such as chronic blood loss, hemolytic anemia, and thalassemia.
* Clinical and/or laboratory evidence of hepatic, renal, cardiovascular abnormalities.
* History of peptic disorders.
* Esophagitis
* Hiatal hernia
* Malabsorption syndrome

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 399 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Treatment of Anemia | 6 months
  Efficacy of lactoferrin alone and lactoferrin with iron for treatment of iron deficiency anemia during 3rd trimester of pregnancy by measuring the hemoglobin level before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali Nasr, Professor, Study Chair — Al-Azhar University, Faculty of medicine, Assuit.; Medhat kamel fathy, Lecturer, Study Director — Al-Azhar University, Faculty of medicine, Assuit.
Locations (1):
- Al-Azhar University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No